CLINICAL TRIAL: NCT04632420
Title: Evaluation of Headache and Childbirth in a Chronic Pain Population
Status: Completed | Type: Observational
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Pamela Flood, Professor, Stanford University
Other Study IDs: 52732b
Record Dates: First submitted 2020-10-30; First posted 2020-11-17 (Actual); Last update posted 2023-04-11 (Actual); Status verified 2023-04

CONDITIONS: Headache
MeSH Terms: conditions — Headache

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Women with child birth: Women attending chronic pain clinic who have previously experienced childbirth
- Women without childbirth: Women attending chronic pain clinic who have not previously experienced childbirth

SUMMARY:
Headache and backache are common symptoms following childbirth. The incidence of these symptoms have been shown to increase during the postpartum period between 5 to 12 months following delivery. By 12 months postpartum up to 45% and 65% of women experience headache and backache, respectively. While studies have reported headache and backache as frequently persistent symptoms beyond the first year postpartum, few studies have specifically interrogated women seeking specialist pain physician input or identified predisposing risk factors. Finally there is little known about typically described pain characteristics of women who suffer with chronic postpartum headache and backache. We aim to compare the prevalence of chronic headache in women that have versus have not experienced childbirth.

ELIGIBILITY:
Inclusion Criteria:

* Women greater than 18 years old
* Agreeing to be contacted for research purposes.
* Able to read and understand English who have had agreed to be contacted with a valid email address

Exclusion Criteria:

* Self identified as non-female
* Age <18 years old.
* Women without computer or electronic device access or valid email address and women who did not respond

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Women who went to the pain clinic and fulfill the inclusion and exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 1112 (Actual)
Dates: Start 2019-09-13 (Actual); Primary Completion 2020-02-26 (Actual); Study Completion 2020-02-26 (Actual)

PRIMARY OUTCOMES:
Prevalence of chronic headache | 10 minute questionnaire
  Percentage of patients with chronic headache in women who have given birth and who have not given birth

SECONDARY OUTCOMES:
Severity of headache | 10 minute questionnaire
  1 to 10 scale. 1 is almost no pain, 10 is worst pain imaginable
Frequency of worst headache | 10 minute questionnaire
  How many days per month did patients have worst headaches
Age of onset of headache | 10 minute questionnaire
  Age of onset of headache
Postpartum headache | 10 minute questionnaire
  Percentage of headache in the postpartum period in women who have given birth
Predictors for postpartum headache | 10 minute questionnaire
  Association between demographics/headache characteristics/predisposing risk factors and postpartum headache
Risk factors for developing acute or acutely worsened headache within 5 days of delivery | 10 minute questionnaire
  Association between demographic, obstetric or anesthesia related factors and acute or acutely worsened headache within 5 days of delivery

CONTACTS AND LOCATIONS:
Locations (1):
- Stanford University, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No